CLINICAL TRIAL: NCT06928779
Title: An Open-Label, Single-Dose, Adaptive Design Study to Evaluate the Effects of Hepatic Impairment on the Pharmacokinetics of Dazucorilant
Brief Title: Effects of Hepatic Impairment on the Pharmacokinetics of Dazucorilant
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Corcept Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CORT113176-657
Record Dates: First submitted 2025-04-08; First posted 2025-04-15 (Actual); Last update posted 2025-04-15 (Actual); Status verified 2025-04

CONDITIONS: Hepatic Impairment
MeSH Terms: interventions — CORT113176

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Moderate Hepatic Impairment (Experimental): On Day 1, each participant with moderate hepatic impairment will receive a single oral dose of dazucorilant 300 mg.
  Interventions: Drug: Dazucorilant
- Matched Healthy Participants (Experimental): Healthy participants will be matched to those with moderate hepatic impairment as to gender, age (± 10 years of the mean), and weight (± 20% of the mean). On Day 1, each healthy participant will receive a single oral dose of dazucorilant 300 mg.
  Interventions: Drug: Dazucorilant
- Mild Hepatic Impairment (Experimental): On Day 1, each participant with mild hepatic impairment will receive a single oral dose of dazucorilant 300 mg. This arm may be enrolled after review of interim PK evaluation of the effects of moderate hepatic impairment.
  Interventions: Drug: Dazucorilant

INTERVENTIONS:
Drug: Dazucorilant — Dazucorilant 300 mg (4 X 75 mg) soft gelatin capsules for oral administration
  Other Names: CORT113176

SUMMARY:
This study will compare the pharmacokinetics (PK) of dazucorilant (CORT113176) between participants with normal hepatic function and participants with hepatic impairment.

DETAILED DESCRIPTION:
Initially, participants with moderate hepatic impairment and healthy control participants matched as to gender, age, and weight will be enrolled. After completing screening assessments, participants will receive a single dose of dazucorilant followed by an observation period of 7 days. Based on the observed effect of moderate hepatic impairment on the dazucorilant PK profile, and review of safety data, a group of participants with mild hepatic impairment, matched to the enrolled healthy control participants, may be enrolled to evaluate the effects of mild hepatic impairment on dazucorilant PK.

ELIGIBILITY:
Inclusion Criteria:

* A non-smoker (no use of tobacco or nicotine products within 3 months prior to Screening) or light smokers (no more than 5 cigarettes/day or nicotine equivalent)
* Has body mass index (BMI) ≥18.0 and ≤32 kg/m^2 and body weight ≥50.0 kg
* Female participants (except for post-menopausal and surgically sterile women) who are sexually active with a non-sterile male partner must be willing to use 1 of the acceptable contraceptive methods described in the protocol throughout the study and for 90 days after study drug administration
* Female participants of non-childbearing potential must be post-menopausal or surgically sterile
* Male participants who are not vasectomized at least 6 months prior to study drug administration and who are sexually active with a non-sterile female partner must be willing to use 1 of the acceptable contraceptive methods described in the protocol from dosing until at least 90 days after study drug administration
* Male participants must be willing not to donate sperm until 90 days following the administration of the study drug
* Has estimated glomerular filtration rate ≥60 mL/min/1.73 m^2 at Screening
* Is able to understand the study procedures, agree to abide by the study restrictions, and provide signed informed consent to participate in the study.

Additional Inclusion Criteria for Healthy Control Group Participants Only:

* Healthy as defined by: a) on a population basis, matched to participants with moderate hepatic impairment according to gender, age (±10 years), and weight (±20%); b) BMI ≥18.0 and ≤32 kg/m^2; c) the absence of clinically significant history of neurological, endocrine, cardiovascular, pulmonary, hematological, immunologic, psychiatric, gastrointestinal, renal, hepatic (including cholecystectomy), and metabolic disease; and d) no clinically significant deviation for laboratory tests results.

Additional Inclusion Criteria for Participants with Hepatic Impairment Only:

* Documented parenchymal hepatic disease evidenced by, e.g., ultrasonography, computed tomography (CT), magnetic resonance imaging (MRI), Fibroscan, or biopsy
* Chronic (≥6 months) hepatic impairment (of any etiology) that has been clinically stable for at least 1 month prior to Screening as determined by the Principal Investigator (PI). Participants must also remain stable throughout the screening period
* Has hepatic impairment as assessed by a Child-Pugh classification score: Mild (5-6 points) or Moderate (7-9 points) according to hepatic function group
* Has normal or non-clinically significant findings at physical examination and normal limits or non-clinically significant deviations in clinical laboratory evaluations with the exception of findings that in the opinion of the PI are consistent with participant's hepatic impairment or other stable chronic medical condition
* Has a stable drug regimen for 14 days prior to study drug administration. Medications are allowed if they are essential for the management of hepatic impairment and the treatment of concomitant stable medical conditions for the hepatically impaired participants.

Exclusion Criteria:

* Clinically significant illness or surgery within 4 weeks prior to dosing
* Gastrointestinal surgery that interferes with physiological absorption and motility (e.g. gastric bypass, duodenectomy) or gastric bands
* Clinically significant history or presence of any gastrointestinal pathology (e.g. chronic diarrhea, inflammatory bowel diseases), unresolved gastrointestinal symptoms (e.g. diarrhea, vomiting) that can interfere with drug absorption
* History of suicidal tendency, disposition to seizures, state of confusion, or clinically relevant psychiatric diseases
* Has any medical condition that could be aggravated by glucocorticoid antagonism, such as autoimmune disease or rheumatic disease
* Has clinically significant ECG or vital sign abnormalities at Screening
* Has acute viral hepatitis in the 6 calendar months before the administration of the study drug
* Has Gilbert's syndrome, an inherited (genetic) liver disorder that affects the body's ability to process bilirubin
* Has uncontrolled hyperlipidemia (abnormally high levels of lipids in the blood), which include cholesterol and triglycerides) as judged by the PI
* History of significant drug abuse within 1 year prior to Screening or recreational use of soft drugs (such as marijuana) within 1 month, or hard drugs (such as cocaine, phencyclidine [PCP], crack, opioid derivatives including heroin, and amphetamine derivatives) within 3 months prior to Screening, unless for hepatic impaired participants only, the participant uses any of these drugs as prescriptions
* History of significant alcohol abuse within 6 months prior to Screening or regular use of alcohol within 6 months prior to the screening visit (more than 14 units of alcohol per week [1 unit = 150 mL of wine, 360 mL of beer, or 45 mL of 40% alcohol])
* Donation of plasma within 7 days prior to dosing. Donation or loss of blood (excluding volume drawn at Screening or menses) of 50 mL to 499 mL of blood within 30 days, or more than 499 mL within 56 days prior to the dosing
* Female participants with a positive pregnancy test at Screening or Day -1
* Has a positive alcohol (breath or urine) test at Screening or Day -1
* Has a history of clinically significant hypersensitivity to dazucorilant, other related drugs, or any of the ingredients or excipients of the study drug
* Previous participation in a study with dazucorilant administration
* Participated in a clinical research study involving the administration of an investigational or marketed drug or device within 30 days prior to dosing, administration of a biological product in the context of a clinical research study within 90 days prior to dosing, or concomitant participation in an investigational study involving no drug or device
* Participants who have taken a) oral, parenteral, depot or intra-articular glucocorticoids within 12 calendar months prior to study drug administration or b) intranasal, topical, or inhaled glucocorticoids within 2 weeks (or 5 half-lives, if longer) prior to study drug administration
* Use of any drugs, herbal products, or other substances known to induce or inhibit hepatic drug metabolism (including St. John's wort) within 30 days prior to study drug administration
* Male participants (including men who have had a vasectomy) with a pregnant or lactating partner
* Breast-feeding female participants
* Has inability or difficulty to swallow soft gelatin capsules
* Has inability to be venipunctured and/or tolerate catheter venous access
* Is an employee or family member of a contract research organization or Sponsor
* Any reason which, in the opinion of the PI, would prevent the participant from participating in the study.

Additional Exclusion Criteria for Healthy Control Group Participants Only:

* Has previously documented parenchymal hepatic disease evidenced by, for example, ultrasonography, CT, MRI, or biopsy. There is no requirement that control group participants have previously undergone any of these investigations, but results of any that have been performed must be negative
* Has any clinically significant abnormality at physical examination, clinically significant abnormal laboratory test results, or positive test for hepatitis B surface antigen, hepatitis C virus (HCV), or human immunodeficiency virus (HIV) at Screening
* Participants using medication other than topical products without significant systemic absorption: a) prescription medication within 14 days prior to the administration of study drug, b) over-the-counter (OTC) products and natural health products (including herbal remedies, homeopathic and traditional medicines, probiotics, food supplements such as vitamins, minerals, amino acids, essential fatty acids, and protein supplements used in sports) within 7 days prior to dosing, with the exception of the occasional use of acetaminophen (up to 2 g daily), and c) a depot injection or an implant of any drug within 3 months prior to the administration of study drug
* Participants with a positive urine drug screen at Screening or check-in.

Additional Exclusion Criteria for Participants with Hepatic Impairment Only:

* Has clinically significant unstable medical conditions or clinically significant acute exacerbation of hepatic disease within 30 days of study drug administration in the opinion of the PI
* Has clinically significant abnormalities of laboratory, ECG, or clinical data that would preclude participation in the study in the opinion of the PI
* Has presence of chronic kidney disease
* Has presence of hepatocellular carcinoma or acute hepatic disease from infection or drug toxicity
* Has presence of clinically significant history of lactic acidosis and severe hepatomegaly with steatosis
* Has presence of active stage 2, 3, or stage 4 hepatic encephalopathy
* Has evidence of severe ascites at PI's discretion
* Has Type 1 or uncontrolled Type 2 diabetes (decompensated diabetes, glycated hemoglobin HbA1c >10 %)
* Has presence of surgically-created or transjugular intrahepatic portal systemic shunts
* Has a positive test for HIV
* Has a positive drug screen at Screening or check-in. Participants who have a positive drug screen due to prescription drug use will be allowed if approved by the PI
* Use of prohibited concomitant medication. At the discretion of the PI and Medical Monitor and with agreement of the participant's usual physician if applicable, a suitable substitute medication may be prescribed to replace the prohibited medication
* Has history or clinical evidence of hepatic decompensation
* Has history of liver transplant, or current placement on a liver transplant list
* Use of medications for the timeframes specified below, with the exception of medications exempted by the PI on a case-by-case basis because they are judged unlikely to affect the PK profile of the study drug or participant safety: a) prescription medications from 14 days prior to dosing (exceptions apply), or b) OTC and natural health products from 7 days prior to dosing unless a hepatic participant is taking such products for their routine care, with the exception of the occasional use of acetaminophen.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2024-10-08 (Actual); Primary Completion 2024-12-09 (Actual); Study Completion 2024-12-09 (Actual)

PRIMARY OUTCOMES:
Area under the concentration-time curve from time zero to the last non-zero concentration (AUC0-t) of dazucorilant | Predose and at serial timepoints up to 24 hours after dosing, and at 48, 72, 96, 120, and 144 hours after dosing
Area under the concentration-time curve from time zero to infinity (extrapolated) (AUC0-inf) of dazucorilant | Predose and at serial timepoints up to 24 hours after dosing, and at 48, 72, 96, 120, and 144 hours after dosing
Maximum observed concentration (Cmax) of dazucorilant | Predose and at serial timepoints up to 24 hours after dosing, and at 48, 72, 96, 120, and 144 hours after dosing
Time to maximum concentration (Tmax) of dazucorilant | Predose and at serial timepoints up to 24 hours after dosing, and at 48, 72, 96, 120, and 144 hours after dosing
Apparent clearance (Cl/F) of dazucorilant | Predose and at serial timepoints up to 24 hours after dosing, and at 48, 72, 96, 120, and 144 hours after dosing

SECONDARY OUTCOMES:
Number of participants with 1 or more adverse events | Up to Day 7
Number of participants with 1 or more clinically significant abnormal vital signs | Up to Day 7
Number of participants with 1 or more clinically significant abnormal electrocardiogram (ECG) result | Up to Day 7
Number of participants with 1 or more clinically significant abnormal clinical laboratory result | Up to Day 7
Number of participants with 1 or more clinically significant abnormal physical examination result | Up to Day 7

CONTACTS AND LOCATIONS:
Overall Officials: Jeevan Kunta, PhD, Study Director — Corcept Therapeutics
Locations (2):
- United States (2):
  - Site 2, Rialto, California
  - Site 1, Miami, Florida

IPD SHARING:
Plan to Share IPD: No